CLINICAL TRIAL: NCT03142893
Title: Hormonal Mechanisms of Sleep Restriction - Axis Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter y. Liu (Other)
Responsible Party: Sponsor-Investigator, Peter y. Liu, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 30068-01A
Record Dates: First submitted 2017-04-11; First posted 2017-05-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sleep Restriction
Keywords: testosterone; cortisol
MeSH Terms: interventions — Ketoconazole; ganirelix; Dexamethasone; Calcium Dobesilate; Luteinizing Hormone, beta Subunit; Hydrocortisone; hydrocortisone hemisuccinate; Gonadotropin-Releasing Hormone; Corticotropin-Releasing Hormone; corticorelin ovine; Saline Solution; Injections

STUDY DESIGN:
Intervention Model Description: Blood is sampled every 10 minutes from 4PM to 9PM for future mathematical deconvolution in order to determine hormone pulse characteristics in response to the clamp conditions. These values are the primary endpoints.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 3 of the 4 conditions are masked by use of identical injections and pills. However one condition (adrenal testis) is not masked. Hence the study is partially masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control Condition (Experimental): 8 am - Saline Solution for Injection 10 am - Placebo oral capsule
  1 pm - Saline Solution for Injection 4 pm - Placebo oral capsule & start hourly blood sampling 7 pm - Gonadorelin (GnRH) and Corticorelin (CRH) injections 9 pm - Saline Solution for Injection & last blood sample
  Interventions: Drug: Gonadorelin; Drug: Corticorelin; Drug: Placebo oral capsule; Drug: Saline Solution; Drug: Saline Solution for Injection
- Hypothalamic Condition (Experimental): 8 am - Ganirelix 10 am - Placebo oral capsule
  1 pm - Dexamethasone injection 4 pm - Placebo oral capsule and start of hourly blood sampling 7 pm - GnRH and CRH injections 9 pm - Saline Solution for Injection and last sample of blood taken
  Interventions: Drug: Ganirelix; Drug: Dexamethasone Injection; Drug: Gonadorelin; Drug: Corticorelin; Drug: Placebo oral capsule; Drug: Saline Solution for Injection
- Pituitary Condition (Experimental): 8am - Saline Solution for Injection 10am - Ketoconazole Pill
  1pm - Saline Solution for Injection 4pm - Ketoconazole Pill & start of hourly blood sampling 7pm - GnRH and CRH 9pm - Hydrocortisone Injection & last blood sample
  Interventions: Drug: Ketoconazole Pill; Drug: Hydrocortisone Injection; Drug: Gonadorelin; Drug: Corticorelin; Drug: Saline Solution
- Adrenal/Testis Condition (Experimental): 10pm - Ganirelix Injection & Dexamethasone Pills (night before) 8am - start of hourly blood sampling 10am - Dexamethasone Pills 11am - last hourly blood sample taken 11:30am - start of blood sampling every 10 minutes
  1pm - Recombinant Human Luteinizing Hormone (rhLH) Injection 3pm - rhLH Injection 5pm - rhLH Injection 5pm - Cosyntropin Injectable product 7pm - GnRH and CRH Injections 9pm - last blood sample taken
  Interventions: Drug: Ganirelix; Drug: Dexamethasone; Drug: Cosyntropin Injectable Product; Drug: Recombinant Human Luteinizing Hormone; Drug: Gonadorelin; Drug: Corticorelin

INTERVENTIONS:
Drug: Ketoconazole Pill — Ketoconazole pill is taken 4 times per Inpatient Stay
  Other Names: Nizoral
  Arms: Pituitary Condition
Drug: Ganirelix — Ganirelix subcutaneous injection is administered twice per Inpatient Stay
  Arms: Adrenal/Testis Condition; Hypothalamic Condition
Drug: Dexamethasone — Dexamethasone Pills is taken twice per Inpatient Stay
  Arms: Adrenal/Testis Condition
Drug: Dexamethasone Injection — Dexamethasone IV injection is given twice per Inpatient Stay
  Arms: Hypothalamic Condition
Drug: Cosyntropin Injectable Product — cosyntropin injection is given twice per Inpatient Stay
  Arms: Adrenal/Testis Condition
Drug: Recombinant Human Luteinizing Hormone — Leutinizing-Releasing Hormone is given 6 IV infusion pulses per Inpatient Visit
  Other Names: Luveris
  Arms: Adrenal/Testis Condition
Drug: Hydrocortisone Injection — Hydrocortisone IV push is given twice per Inpatient Visit
  Other Names: solu-cortef
  Arms: Pituitary Condition
Drug: Gonadorelin — Gonadorelin IV injection is given twice per Inpatient Stay
  Other Names: Lutrepulse
Drug: Corticorelin — Corticorelin IV injection is given twice per Inpatient Stay
  Other Names: Acthrel
Drug: Placebo oral capsule — Placebo for ketoconazole are given 4 times per Inpatient Stay
  Arms: Control Condition; Hypothalamic Condition
Drug: Saline Solution — Saline Solution (Placebo) for Dexamethasone IV injection or hydrocortisone IV injection given up to four times per Inpatient Stay
  Arms: Control Condition; Pituitary Condition
Drug: Saline Solution for Injection — Saline Solution (placebo) for ganirelix subcutaneous injection
  Arms: Control Condition; Hypothalamic Condition

SUMMARY:
The purpose of this study is to 1) determine how hypothalamic-pituitary-adrenal axis (HPA axis) activation occurs with sleep restriction 2) evaluate how hypothalamic-pituitary-gonadal axis (HPG axis) deactivation occurs with sleep restriction. The investigator will also examine the cognitive function associated with sleep restriction, including food intake and food cravings.

DETAILED DESCRIPTION:
Sleep restriction increases evening cortisol and decreases testosterone. These are the main catabolic and anabolic hormones in men, respectively. This catabolic-anabolic imbalance likely leads to metabolic and reproductive ill-health. The hypothalamic-pituitary-end organ (adrenal or testis) mechanisms that must underpin these changes are unknown. This study will administer drugs to clamp the function of each of these nodes to determine the regulatory changes that have occurred with sleep restriction. Even though the study is randomized order in design, the main comparison is before and after sleep restriction under each of these clamp conditions. Participants are admitted to the chronobiology laboratory where they are given 1 night of 10 hours sleep opportunity, followed by 4 nights of 4 hours sleep opportunity. Up to 80 participants (assuming twenty different participant for each of the 4 clamp conditions) can be enrolled. However, participants will be allowed an opportunity to be randomized to all 4 conditions so that as few as 20 participants may be required. Urn randomization will be used to ensure that 20 different participants are involved in each of the 4 conditions.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 22-45 years
* Willingness to provide written informed consent
* Stable weight over preceding 6 weeks
* Body Mass index (BMI) 20-28 kg/m2

Exclusion Criteria:

* Unable or unwilling to provide IRB (Internal Review Board)-approved informed consent
* Clinical disorders and/or illnesses
* Current medical or drug treatment, as assessed by questionnaire
* History of brain injury or of learning disability - Vision or hearing impairment unless corrected back to normal
* Anemia (Hct <38%)
* History of psychiatric illness
* Clinically significant abnormalities in blood and urine, and free of traces of drugs
* Other endocrine abnormalities including hypothyroidism or adrenal failure; primary gonadal disease as indicated by serum LH (luteinizing hormone) or FSH (follicle stimulating hormone) concentration >10 or >15 IU/L, respectively, hyperprolactinemia indicated by prolactin >25ug/L
* Type 2 Diabetes (HgbA1C)
* Current smoker
* Recent or concurrent drug or alcohol abuse
* Blood donation in previous eight weeks
* Travel across time zones within one month of entering the study
* Sleep or circadian disorder
* Shift work within three months of entering the study
* Irregular bedtimes (not between 6 and 10 hours in duration)
* Unoperated obstructive uropathy, recurrent prostatitis, indeterminate prostatic nodularity, Hx or Suspicion of cancer of the prostate gland or PSA (prostate-specific antigen) >4ng/ml
* Previous adverse reaction to sleep deprivation or any of the drugs to be administered
* Concurrent participation in another research study

Ages: 22 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Average Blood Cortisol Concentration | 5 days
  Cortisol is measured in blood every 10 minutes for a 5 hour period, at the beginning and at the end of 4 nights of sleep restriction. The average cortisol is the parameter of interest.
Average Blood Testosterone Concentration | 5 days
  Testosterone is measured in blood every 10 minutes for a 5 hour period, at the beginning and at the end of 4 nights of sleep restriction. The average cortisol is the parameter of interest.

SECONDARY OUTCOMES:
Peak Blood Cortisol Concentration | 5 days
  This is the single maximal blood cortisol concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Peak Blood Testosterone Concentration | 5 days
  This is the single maximal blood testosterone concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Trough Blood Cortisol Concentration | 5 days
  This is the single minimal blood cortisol concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Trough Blood Testosterone Concentration | 5 days
  This is the single minimal blood testosterone concentration that is measured during the entire 5 hour period, at the beginning and at the end of 4 nights of sleep restriction.
Reaction time on Psychomotor Vigilance Task | 5 days
  This is measured by lapses in attention. As the person becomes more sleepy, there are more lapses (reaction time >500 ms), at the beginning and at the end of 4 nights of sleep restriction.
Karolinska Sleepiness Scale | 5 days
  Measures how sleepy participants are using a scale of 1 (extremely alert) through 9. This scale will be used to assess changes in sleepiness throughout the day and through 4 nights of sleep restriction.
Two card gambling task | 5 days
  Computerized neurobehavioral testing to determine how 4 nights of sleep restriction affects participants' decision making. The end point is discriminability index, d'.
Modified Sternberg working memory test | 5 days
  Computerized neurobehavioral testing to determine how 4 nights of sleep restriction affects reaction time and accuracy.
Caloric Intake | 5 days
  The food given to participants is weighed. The amount that is not consumed is also weighed. The difference in weight is the amount of calories consumed.
Hunger Scale | 5 days
  Hunger scale using Flint visual analogue scale to assess how 4 nights of sleep restriction affects participants' appetite.
Food Cravings | 5 days
  Food cravings is measured using Food Cravings Index scale to assess which food groups participants have cravings for and how their cravings change during 4 nights of sleep restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MD, PhD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No